CLINICAL TRIAL: NCT01669980
Title: A Multicenter, Randomized, Observer-Blinded, Active-Controlled Study Evaluating the Safety, Tolerability, Pharmacokinetics, and Efficacy of Ceftaroline Versus Ceftriaxone Plus Vancomycin in Pediatric Subjects With Complicated Community-acquired Bacterial Pneumonia (CABP)
Brief Title: Safety and Efficacy Study of Ceftaroline Versus a Comparator in Pediatric Subjects With Complicated Community Acquired Pneumonia (CABP)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P903-24
Record Dates: First submitted 2012-08-17; First posted 2012-08-21 (Estimated); Last update posted 2015-11-02 (Estimated); Status verified 2015-10

CONDITIONS: Infections; Pneumonia
Keywords: Infections; Pediatrics; Teflaro; Ceftriaxone; cephalosporin; Vancomycin; Clindamycin; Amoxicillin Clavulanate; Linezolid; MRSA; pneumonia
MeSH Terms: conditions — Infections; Pneumonia | interventions — Ceftaroline; Ceftriaxone; Vancomycin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ceftaroline fosamil (Experimental)
  Interventions: Drug: Ceftaroline fosamil
- IV Ceftriaxone and Vancomycin (Active Comparator)
  Interventions: Drug: IV Ceftriaxone and Vancomycin

INTERVENTIONS:
Drug: Ceftaroline fosamil — * Subjects ≥ 6 months: IV ceftaroline fosamil 15 mg/kg (or 600 mg if > 40 kg) infused over 120 (± 10) minutes q8h (± 1 hour)
  * Subjects < 6 months: IV ceftaroline fosamil 10 mg/kg infused over 120 (± 10) minutes q8h (± 1 hour)
  Optional Oral Switch:
  * PO amoxicillin clavulanate 45 to 90 mg/kg/day divided q12h
  * PO clindamycin 13 mg/kg/dose
  * PO linezolid 600 mg q12h (Cohort 1) or 10 mg/kg q8h
  Other Names: Teflaro; PPI-0903; TAK-599; TAK599; PPI0903
  Arms: Ceftaroline fosamil
Drug: IV Ceftriaxone and Vancomycin — * IV ceftriaxone 75 mg/kg/day (up to 4 g/day) divided equally every 12 hours (q12h) (± 2 hours) infused over 30 (± 10) minutes AND
  * IV vancomycin 15 mg/kg every 6 hours (q6h) (± 1 hour) infused over at least 60 minutes.
  Optional Oral Switch:
  * PO amoxicillin clavulanate 45 to 90 mg/kg/day divided q12h
  * PO clindamycin 13 mg/kg/dose
  * PO linezolid 600 mg q12h (Cohort 1) or 10 mg/kg q8h
  Arms: IV Ceftriaxone and Vancomycin

SUMMARY:
This is a study of safety and effectiveness of ceftaroline fosamil in children with Complicated Community-acquired Pneumonia receiving antibiotic therapy in the hospital.

DETAILED DESCRIPTION:
To evaluate safety, effectiveness, pharmacokinetics and tolerance of ceftaroline fosamil in pediatric subjects ages 2 months to < 18 years who are initially hospitalized with Complicated Community Acquired Bacterial Pneumonia (CABP) at high risk of infection due to methicillin-resistant Staphylococcus aureus (MRSA)

ELIGIBILITY:
Inclusion Criteria:

* Presence of CABP warranting 3 days of initial hospitalization
* Confirmed presence of indicators of complicated CABP

Exclusion Criteria:

* Hypersensitivity or allergic reaction to vancomycin or any β-lactam antimicrobial
* Confirmed or suspected infection with a pathogen known to be resistant to IV study drugs or known infection at baseline with a sole atypical organism
* Confirmed or suspected respiratory tract infection attributable to sources other than community acquired bacterial pneumonia
* Non-infectious causes of pulmonary infiltrates

Ages: 2 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2012-10; Primary Completion 2014-05 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety and tolerability of ceftaroline versus ceftriaxone plus vancomycin in pediatric subjects ages 2 months to < 18 years with complicated community-acquired bacterial pneumonia (CABP) | between 1 and 57 days
  Evaluate the safety and tolerability of IV administered ceftaroline fosamil in children with complicated CABP. Summaries of patient AEs, SAEs, deaths, discontinuations due to AEs, laboratory evaluations (hematology studies, comprehensive and metabolic panel), and vital signs will be provided for each treatment group.

SECONDARY OUTCOMES:
To evaluate the efficacy of ceftaroline versus ceftriaxone plus vancomycin in pediatric subjects with complicated CABP at high risk of infection due to methicillin-resistant Staphylococcus aureus (MRSA). | between 4 and 57 days
  Evaluate the efficacy of ceftaroline versus ceftriaxone plus vancomycin in pediatric subjects with complicated CABP at high risk of infection due to methicillin-resistant Staphylococcus aureus (MRSA) by assessing clinical stability of the subject at study day 4 and clinical outcome at End of IV, End of Treatment and Test of Cure.
Evaluate the pharmacokinetics of ceftaroline in pediatric subjects with complicated CABP at high risk of infection due to methicillin-resistant Staphylococcus aureus (MRSA) | between 4 and 57 days
  Analyze concentrations of ceftaroline, ceftaroline fosamil (prodrug), and ceftaroline M-1 (inactive metabolite) in plasma, and, if available, in cerebrospinal fluid (CSF, if collected as part of standard of care)

CONTACTS AND LOCATIONS:
Locations (21):
- United States (13):
  - Investigational Site, Long Beach, California
  - Oakland, California
  - Investigational Site, Orange County, California
  - Investigational Site, San Diego, California
  - Investigational Site, Boston, Massachusetts
  - Investigational Site, Cleveland, Ohio
  - Investigational Site, Toledo, Ohio
  - Investigational Site, Pittsburgh, Pennsylvania
  - Investigational Site, Memphis, Tennessee
  - Houston, Texas
  - Salt Lake City, Utah
  - Investigational Site, Norfolk, Virginia
  - Investigational Site, Morgantown, West Virginia
- Investigative Site, Buenos Aires, Argentina
- Georgia (3):
  - Investigational Site 1, Tbilisi
  - Investigational Site 2, Tbilisi
  - Investigational Site 3, Tbilisi
- Ukraine (4):
  - Investigational Site, Donetsk
  - Investigational Site, Ivano-Frankivsk
  - Investigational Site, Kryvyi Rih
  - Investigational Site, Kyiv

REFERENCES:
- See also: Sponsor Homepage — http://www.cerexa.com